CLINICAL TRIAL: NCT06762106
Title: Effect of Shockwave Therapy on Low Back Pain in Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deraya University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: physio 12 24
Record Dates: First submitted 2024-12-30; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Dysmenorrhea; Back Pain Lower Back
Keywords: dysmenorrhea; lower back pain; shock wave
MeSH Terms: conditions — Dysmenorrhea; Low Back Pain | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hot back group (Active Comparator): 30 subjects were treated by hot back in the first 3 days of the menstrual cycle (follicular phase) for three consecutive menstrual cycles
  Interventions: Radiation: hot back
- shock wave and hot back group (Experimental): 30 subjects were treated by hot back and shockwave therapy in the first 3 days of the menstrual cycle (follicular phase) for three consecutive menstrual cycles
  Interventions: Radiation: shockwave therapy

INTERVENTIONS:
Radiation: shockwave therapy — solid unite made with metal frame and case
  Arms: shock wave and hot back group
Radiation: hot back — thermal hot back
  Arms: Hot back group

SUMMARY:
Primary dysmenorrhea (PD), defined as menstrual pain without any structural lesions, usually begins shortly before or immediately after the onset of the menstrual cycle and commonly lasts for 48 to 72 hour

DETAILED DESCRIPTION:
Dysmenorrhea is one of the most common gynecological conditions in women. Primary dysmenorrhea (PD), defined as menstrual pain without any structural lesions, usually begins shortly before or immediately after the onset of the menstrual cycle and commonly lasts for 48 to 72 hour. It is accompanied by general symptoms, such as nausea and vomiting, malaise, weakness, lower backache, and diarrhea. In ovulatory cycles, women secrete high levels of or have increased sensitivity to prostaglandins. These prostaglandins may stimulate myometrial contractions and sensitize pain fibers, and thus induce pelvic pain.

Females of reproductive age often suffer from dysmenorrhea, a painful condition. Despite dysmenorrhea being generally considered a benign condition, a significant disability can result from it. Researchers suggest that dysmenorrhea has been linked to migraines, headaches, and fibromyalgia, among other painful disorders. The authors reported further evidence that dysmenorrhea can alter noxious sensory processing.

Primary dysmenorrhea usually begins six to 12 months after menarche and is characterized by spasmodic cramping pain in the lower abdomen that can radiate to the lower back and anterior or inner thighs. The pain usually has a clear temporal pattern: it begins a few hours before or at the start of menstruation, is most intense at onset, gradually waning over two to three days.

The purpose of this study was to investigate the effectiveness shockwave therapy on low back pain in primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Their ages ranged from 18 to 30 years.
* Their BMI were not exceeding 29 Kg/m2.
* All patients were clinically diagnosed as low back pain during Primary Dysmenorrhea according to the Primary Dysmenorrhea Consensus Guideline

Exclusion Criteria:

* Any known chronic disease (such as cardiovascular or renal diseases) or secondary dysmenorrhea.
* Being pregnant or planning to get pregnant any time during the trial.
* Having received other treatments for PD in the past half year.
* Irregular menstrual cycles.
* Mental or neurological disorder

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — as menstruation is found only in females
Enrollment: 60 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-03-02 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Pain assessment | every month for three menstrual cycle
  VAS scoring method. 0 is the least while 10 is the highest

CONTACTS AND LOCATIONS:
Locations (1):
- Minia, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No